CLINICAL TRIAL: NCT01542333
Title: Biological Analysis of Ethnic Variations in Wilms Tumor
Brief Title: Studying Biomarkers in Samples From Younger Patients With Wilms Tumor
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN12B2; COG-AREN12B2 (Other: Children's Oncology Group); CDR0000726713 (Other: Clinical trials.gov); AREN12B2 (Other: Children's Oncology Group); NCI-2012-00686 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-02-22; First posted 2012-03-02 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Cancer
Keywords: recurrent Wilms tumor and other childhood kidney tumors; stage I Wilms tumor; stage II Wilms tumor; stage III Wilms tumor; stage IV Wilms tumor; stage V Wilms tumor
MeSH Terms: conditions — Kidney Neoplasms; Wilms Tumor | interventions — Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction; Blotting, Western; Immunohistochemistry; Spectrum Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: proteomic profiling
Genetic: reverse transcriptase-polymerase chain reaction
Genetic: western blotting
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: spectroscopy

SUMMARY:
RATIONALE: Studying samples of tissue and urine from patients with cancer in the laboratory may help doctor learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies biomarkers in samples from younger patients with Wilms tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine a unique molecular "finger print" of primary Wilms tumor arising in ethnically diverse children who are at increased risk to develop this lethal malignancy and subsequently relapse.
* To determine a unique protein "finger print" from the urine of ethnically diverse children who develop Wilms tumor and subsequent relapse.

OUTLINE: Formalin-fixed paraffin-embedded and snap-frozen primary tissue samples, and urine samples collected at the time of diagnosis and before treatment, are analyzed for molecular and protein profile by MALDI-TOF mass spectroscopy, western blotting, immunohistochemistry, and reverse-transcriptase polymerase chain reaction (RT-PCR) assays.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with Wilms tumor
* Specimens from African-American and from Caucasian children
* Specimens from each ethnicity who relapsed
* Specimens from each ethnicity who did NOT relapse

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosed with Wilms tumor
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Molecular "finger print" of primary Wilms tumor in ethnically diverse children
Protein "finger print" from the urine of ethnically diverse children

CONTACTS AND LOCATIONS:
Overall Officials: Harold N. Lovvorn, III, MD, Principal Investigator — Vanderbilt Children's Hospital